CLINICAL TRIAL: NCT03813212
Title: Gray-scale , Colour Doppler Ultrasound and Magnetic Resonance Imaging for Diagnosis of Placenta Accreta
Brief Title: Magnetic Resonance Imaging (MRI ) Versus Ultrasound in Placenta Accreta Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Safaa thabet abd El Aziz Ahmed, Principal investigator, Ain Shams University
Other Study IDs: MRI placenta accreta
Record Dates: First submitted 2018-11-17; First posted 2019-01-23 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Placenta Accreta, Third Trimester
MeSH Terms: conditions — Placenta Accreta | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — Magnetic resonance imaging. Trans-abdominal sonography (TAS) and transvaginal sonography (TVS) will be performed using a 3.5 or 5 MHz transabdominal convex transducer and a 7 MHz trans-vaginal transducer.
  Other Names: Ultrasound

SUMMARY:
This study aim to assess the accuracy of magnetic resonance imaging (MRI) compared to gray-scale and colour Doppler ultrasound (US) for the prenatal diagnosis of placenta accreta.

DETAILED DESCRIPTION:
Placenta accreta occurs when the chorionic villi abnormally invade the myometrium. Based on histopathology it is divided into three grades: placenta accreta (the chorionic villi are in contact with the myometrium), placenta increta (the chorionic villi invade the myometrium), and placenta percreta where the chorionic villi penetrate the uterine serosa. With increasing rate of cesarean delivery, the incidence of both placenta praevia and placenta accreta is steadily increasing in frequency.

Prenatal diagnosis of invasive placentation is associated with a reduced risk of maternal complications as it allows a preplanned treatment of the condition . Gray-scale and colour Doppler ultrasound (US) are valuable tools in the prenatal diagnosis of placenta accreta .However, if the ultrasound ( US ) findings suggest possible percreta or are inconclusive or negative in an at-risk woman, magnetic resonance imaging (MRI) can be useful.

Multiple sonographic findings are seen with placenta accreta such as decrease in myometrial thickness, placenta previa, placental lacunae, abnormal pattern of color Doppler, loss of the retroplacental clear zone and placenta percreta irregularities in wall of urinary bladder ( UB ) have been detected .

The most magnetic resonance imaging characteristic findings seen in placenta accreta are nodular thickening in the dark zone of placenta-uterine interface together with extensions of dark bands through the placenta, outer uterine bulge causing from the mass effect of the placenta and heterogeneous signal intensity of placenta on the T2-weighted HASTE sequences due to large placental lakes and vessels.

ELIGIBILITY:
Inclusion Criteria:

* Haemodynamically stable pregnant women who have the following risk factors for placenta accreta : persistent anterior placenta previa, prior uterine surgery (such as a previous cesarean section, uterine curettage, or myomectomy).
* Maternal age : 20-40 years old.
* BMI : 18-29.9 kg/m2.

Exclusion Criteria:

* Exclusion criteria will be MRI contraindications, cardiac pacemaker, metal objects in the body, and patient's refusal for MRI evaluation.
* Haemodynamically unstable patients.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Haemodynamically stable pregnant women, who attend the antenatal care clinic at Ain Shams University Hospital or are referred from other hospitals for further evaluation. The recruited patients have to fulfill the inclusion criteria,
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Determination of degree of placental invasion | Baseline
  Determination of degree of placental invasion by comparing the results obtained by ultrasound , MRI with the final pathological examination after operation ( the excised part of myometrium with the attached placenta or hysterectomy specimen ).

SECONDARY OUTCOMES:
Change Maternal morbidity and mortality | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine ainshams university, Cairo, Egypt

REFERENCES:
- [Background] Lopes ES, Feitosa FEL, Brazil AV, de Castro JDV, da Costa JIF, Araujo Junior E, Peixoto AB, Carvalho FHC. Assessment of Sensitivity and Specificity of Ultrasound and Magnetic Resonance Imaging in the Diagnosis of Placenta Accreta. Rev Bras Ginecol Obstet. 2019 Jan;41(1):17-23. doi: 10.1055/s-0038-1675803. Epub 2018 Nov 14. PMID 30428490
- [Background] Haunschild C, Yeaton-Massey A, Lyell DJ. Antenatal Management of Placenta Accreta. Clin Obstet Gynecol. 2018 Dec;61(4):766-773. doi: 10.1097/GRF.0000000000000394. PMID 30204620